CLINICAL TRIAL: NCT03918967
Title: A Two-segment Phase I, Randomized, Double-Blind, Placebo-Controlled, Sequential, Ascending Single and Multiple Dose Study to Evaluate Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of CT-G11 and CT-G20 in Healthy Volunteers (Part 1 and Part 2) and Open Label, Balanced, Randomized, Two-period, Two-Sequence Crossover Study to Assess the Effect of Food on the Pharmacokinetics of CT-G20 in Healthy Volunteers (Part 3)
Brief Title: Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of CT-G20 or CT-G11 and Food Effect of CT-G20 in Human Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Celltrion (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: CT-G20 1.1
Record Dates: First submitted 2019-04-09; First posted 2019-04-18 (Actual); Last update posted 2020-06-09 (Actual); Status verified 2020-06

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- CT-G11 (Experimental): CT-G11 Experimental Drug
  Interventions: Drug: CT-G11
- CT-G20 (Experimental): CT-G20 Experimental Drug
  Interventions: Drug: CT-G20
- CT-G11 Placebo (Placebo Comparator)
  Interventions: Drug: CT-G11 Placebo
- CT-G20 Placebo (Placebo Comparator)
  Interventions: Drug: CT-G20 Placebo

INTERVENTIONS:
Drug: CT-G11 — oral tablet of CT-G11 Experimental Drug
  Arms: CT-G11
Drug: CT-G20 — oral tablet of CT-G20 Experimental Drug
  Arms: CT-G20
Drug: CT-G11 Placebo — oral tablet of Placebo
  Arms: CT-G11 Placebo
Drug: CT-G20 Placebo — oral tablet of Placebo
  Arms: CT-G20 Placebo

SUMMARY:
The purpose of this study is to establish safety, tolerability, pharmacokinetics and pharmacodynamics of CT-G20 or CT-11 and to evaluate potential effect of food on pharmacokinetics of CT-G20 in human participants. It will be conducted in three parts, as described below:

* Part I will be a randomized, double-blind, placebo-controlled, sequential, single ascending dose study.
* Part II will be a randomized, double-blind, placebo-controlled, sequential, multiple ascending dose study.
* Part III will be a randomized, open-label, balanced, two-period, two-sequence crossover, food effect study.

ELIGIBILITY:
Inclusion Criteria:

* body mass index (BMI) ≥18.0 and ≤30.0 kg/m2

Exclusion Criteria:

* Clinically significant allergic reactions
* Gastrointestinal, renal, hematological, metabolic, neurologic or pulmonary diseases classified as significant by the Investigator
* Hepatic dysfunction upper limit of normal laboratory range
* Cardiac history or presence
* History or any concomitant active malignancy
* A known infection with human immunodeficiency virus, hepatitis B virus (HBV) or hepatitis C virus (HCV)
* Inherited bleeding diathesis or coagulopathy with the risk of bleeding
* Hemoptysis, thrombotic or hemorrhagic event
* Cerebral vascular accident, transient ischemic attack, or subarachnoid hemorrhage
* History and/or sign/symptoms of abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess
* Lactose intolerance (lactase deficiency) and glucose-galactose malabsorption

Ages: 19 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 72 (Actual)
Dates: Start 2019-04-08 (Actual); Primary Completion 2020-06-06 (Actual); Study Completion 2020-06-06 (Actual)

PRIMARY OUTCOMES:
Incidence of Adverse events including serious Adverse events (Part I, Part II) | 46 days
Food effect as assessed by : PK parameters including Area under the concentration-time curve (AUC) and Maximum observed concentration (Cmax) (Part III) | Up to 48 hours after administration

SECONDARY OUTCOMES:
Safety parameters as assessed by: QT interval of ECG | 17 Days
Safety parameters as assessed by: QTcF of ECG | 17 Days
Safety parameters as assessed by: blood pressure of Vital signs | 17 Days
Safety parameters as assessed by: pulse rate of Vital signs | 17 Days
Safety parameters as assessed by: body temperature of Vital signs | 17 Days
Safety parameters as assessed by: hematology of Clinical laboratory tests | 17 Days
Safety parameters as assessed by: clinical chemistry | 17 Days
PK parameters as assessed by : Area under the concentration-time curve (AUC) | 13 Days
PK parameters as assessed by : Maximum observed concentration (Cmax) | 13 Days
PK parameters as assessed by : Time to Cmax (tmax) | 13 Days
PK parameters as assessed by : Terminal half-life time (t1/2) | 13 Days
PD parameters as assessed by : Left ventricular ejection fraction (LVEF) | 17 Days

CONTACTS AND LOCATIONS:
Overall Officials: In-Jin Jang, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea